CLINICAL TRIAL: NCT03224559
Title: Applying Neuromodulation to Accelerate Training Effects
Acronym: ANeMATE
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment never began.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00001248
Record Dates: First submitted 2017-06-16; First posted 2017-07-21 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Cognition
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sham Stimulation: subject receives minimal transcranial electrical stimulation
  Interventions: Device: Transcranial Electrical Stimulation
- Left Side Stimulation: transcranial electrical stimulation on the left side of the head.
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — Transcranial Electrical Stimulation
  Other Names: XCITE 100 (Pulvinar Neuro)

SUMMARY:
This study seeks to understand at how noninvasive electrical brain stimulation might change how people perform on on tasks requiring concentration and thinking skills.

DETAILED DESCRIPTION:
This study uses noninvasive electrical stimulation delivered through seeks to understand at how noninvasive electrical brain stimulation might change how people perform on on tasks requiring concentration and thinking skills.

ELIGIBILITY:
Inclusion Criteria:

People may participate in the experiment if they have normal or corrected vision, are in good health, and are at least 18 years old.

Exclusion Criteria:

People will be screened and excluded from participation if they are currently ill or if they report any history of seizures, if they lack the capacity to consent or appear to lack capacity to consent, if they have participated in previous thinking skills training or brain stimulation, or if they are currently taking certain substances/medications that might change thinking skills.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, 18-65 years old
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Working memory | Baseline through 2 months
  Working Memory

CONTACTS AND LOCATIONS:
Overall Officials: Angus W MacDonald, PhD, Principal Investigator — University of Minnesota; Joshua E Mervis, BA, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States